CLINICAL TRIAL: NCT05672082
Title: Contribution of [18F]DPA-714 PET for Grading and Exploration of the Inflammatory Microenvironment of Glioma, a Pilot Study
Brief Title: Contribution of [18F]DPA-714 PET for Grading and Exploration of the Inflammatory Microenvironment of Glioma.
Acronym: INFLAGLI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisational difficulties
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-1-58-002
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]DPA-714 PET (Experimental)
  Interventions: Drug: [18F]DPA-714

INTERVENTIONS:
Drug: [18F]DPA-714 — Participant received one injection of 200 MBq of [18F]DPA-714

SUMMARY:
The 18-kDa translocator protein (TSPO) is a mitochondrial protein that is weakly expressed in the healthy brain. However, there is an increase in the expression of TSPO in glial tumors. It is even associated with a higher malignancy and a shorter survival of patients. Among the different TSPO ligands, the most commonly used tracers in PET imaging are [18F]DPA-714 and 18F-GE180. We hypothesize that [18F]DPA-714 PET could improve the current performance for tumor grade definition in vivo, which is a major issue for the therapeutic management of gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Suspicion of an operable diffuse glioma
* Written informed consent (signed)
* Affiliated or beneficiary of a social security plan

Exclusion Criteria:

* Suspicion of grade I glioma
* Surgical urgency (less than 8 days between the suspected diagnosis and surgery)
* Pregnant or breastfeeding woman
* Persons deprived of liberty or under guardianship
* Impossibility to undergo the medical follow-up of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performances of [18F]DPA-714 PET for glioma grading obtained by stereotactic biopsies of glioma | [18F]DPA-714 PET performed up to 30 days before brain surgery
  Sensitivity and specificity of [18F]DPA-714 PET using anatomopathological assessment of biopsies as gold standard

SECONDARY OUTCOMES:
Comparison of [18F]DPA-714 PET quantitative parameters with anatomopathological assessment of the surgery specimen | [18F]DPA-714 PET performed up to 30 days before brain surgery
  Comparison of [18F]DPA-714 PET quantitative parameters with the histological types of gliomas, with the IDH1-mutational status, and the 1p19q codeletion status
Comparison of [18F]DPA-714 PET quantitative parameters with tumor microenvironment | [18F]DPA-714 PET performed up to 30 days before brain surgery
  Comparison of [18F]DPA-714 PET quantitative parameters with the frequency and phenotype of tumor microenvironment different glioma-associated cells

CONTACTS AND LOCATIONS:
Overall Officials: Xavier PALARD NOVELLO, Dr, Principal Investigator — Centre de lutte contre le cancer Eugène Marquis

IPD SHARING:
Plan to Share IPD: No